CLINICAL TRIAL: NCT03428048
Title: NEXUS Registry: An Outcomes Database Which Tracks Patient -Reported Outcomes After Percutaneous Coronary Intervention for Coronary Artery Disease Along With Surgical and Subcutaneous Ablation for the Management of Atrial Fibrillation.
Brief Title: Cardiovascular Innovation & Research Institute 's NEXUS Registry, the Whole is Greater Than the Parts.
Status: Recruiting | Type: Observational
Sponsor: Cardiovascular Innovation and Research Institute (Other)
Collaborators: Valley View Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2015_01
Record Dates: First submitted 2016-03-15; First posted 2018-02-09 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation (AF)
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation | interventions — Radiofrequency Ablation; Cryosurgery; Laser Therapy; Catheter Ablation; Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults diagnosed with paroxysmal and persistent Afib: Adults diagnosed with paroxysmal and persistent Afib who are identified as candidates for an intervention either surgical (epicardial) known as the hybrid approach or an endocardial ablation with either laser, radio frequency or cryoablation energy source.
  Interventions: Procedure: Hybrid procedure; Procedure: Endocardial ablations; Procedure: left atrial appendage occlusion

INTERVENTIONS:
Procedure: Hybrid procedure — Ablation of the posterior aspect of the heart, an area thought to be the origin of chaotic arrhythmias in persistent Afib patients.
  Other Names: modified maze; epicardial ablation
Procedure: Endocardial ablations — ablations occurring inside the heart isolating the pulmonary veins - blocking energy from creating irregular or chaotic heart beats with use of a catheter
  Other Names: radio frequency ablation; cryoablation; laser ablation; percutaneous ablation
Procedure: left atrial appendage occlusion — A procedure to isolate the left atrial appendage of the heart. this anatomic body is the origin of clot formation which can lead to stroke. the clot formation as a result of Afib
  Other Names: left atrial clip; Watchman procedure; lariat procedure

SUMMARY:
Information gathered from the patients via a disease specific questionnaire will be married to data from the National Cardiovascular Data Registry (NCDR®). Details will be continuously analyzed and used to direct quality of care at our center. The institution is categorized as a low-volume institution for percutaneous coronary intervention (PCI) for coronary artery disease treatment as well as surgical and endocardial ablation for the management of atrial fibrillation (Afib). The association between operator volume and quality has primarily focused on rare complications, such as mortality. The aim is to highlight the advantages of receiving care close to home. A benefit of offering the procedures to treat diseases at centers that have lower volumes is to improve patients' outcomes while also providing more convenient access to quality care. The key outcome from the patients' experience is alleviation of their symptoms while increasing function and quality of life. To date, there have been no studies documenting the health status benefits of PCI and surgical / endocardial ablation for coronary artery disease and Afib, respectively with low- volume operators. In this study, the investigators sought to examine the feasibility of implementing patient-reported outcomes into clinical care and to demonstrate evidence of benefits, from patients' perspectives, of receiving treatment by low-volume operators.

DETAILED DESCRIPTION:
This is a prospective cohort, time series analysis of the routine procedures associated with the catheterization and the electrophysiology lab through ten years post intervention. The goal is to demonstrate clinical effectiveness with cardiac service line with low-volume operators. A connection between NCDR with applied clinical research that directs continuous quality improvement goals and objectives is the ideal setting for value-based, quality care. The system of diagnosing, treating and tracking individuals with cardiovascular and pacing disease has many facets which could benefit from continuous quality improvement and outcomes analysis. The proposed Valley View NEXUS outcomes registry will bridge national data to local clinical data. Clinical registries are a methodically sound instrument for measuring and improving performance. Registries are efficacious for surveillance, measuring effectiveness of quality improvement initiatives, identifying determinates of quality of life and function while synergistically increasing the value of health care expenditures with respect to heart disease, stroke, and arrhythmias.

The ADVARRA formerly Schulman Institutional Review Board (IRB) reviewed our protocol, and authorized the study. Once informed consent was obtained, eligible adults scheduled for diagnostic angiography with possible PCI completed a baseline patient reported outcome assessment and again at designated follow-up intervals (six months and annually thereafter for up to ten years). Due to the urgent nature of STEMI- PCI procedures, it was determined that informed consent prior to PCI was prohibitive; however after consideration, the protocol was amended to capture baseline assessments immediately following PCI while the patient 's status was in hospital with use of the Seattle Angina Questionnaire (SAQ) and the Veterans Rand 12-Item Health Survey (VR-12). The SAQ is recognized as a disease specific questionnaire for coronary artery disease. The SAQ is a six item questionnaire that assesses patient's function, symptoms, and satisfaction. A higher score translates to better outcomes. The VR-12 is a twelve item questionnaire used to assess quality of life. A lower score translates to a higher quality of life in relation to a person's health and wellness. Combining data from a disease specific questionnaire, quality of life assessment, and the NCDR's CathPCI® Registry serves as a nexus between big data and the individual patient experience. From January 2015 through December 2017, twenty- two patients have been enrolled. Based on the data from the first six patients to provide scores both at baseline and month six and with a study design to have 90% power to detect a change in the overall SAQ score of 10 points at six months, it was determined 49 patients will need to be enrolled.

The aforementioned methodology will be applied for surgical and endocardial ablations for patients' with Afib. Presently, enrollment is open for Afib patients and data being captured will be analyzed to determine sample size. Patients who receive intervention for management Afib will complete the Atrial Fibrillation Effect on Quality -of-life (AFEQT) Questionnaire and the VR-12. Again the VR-12 is a twelve item questionnaire used to assess quality of life. A lower score translates to a higher quality of life in relation to a person's health and wellness. The AFEQT is recognized as a disease specific questionnaire for Afib. A higher score translates to worse symptoms and limitations in daily function associated with Afib. Combining the outcomes metric with NCDR's Afib Ablation Registry ® allows our institution demonstrative effective outcomes for low-volume operators.

The data validation process applies to both PCI and surgical and/or endocardial ablation and is as follows:

1. Quality Assurance Plan Training for staff that populates both data registries is ongoing. Staff will participate in the NCDR® applicable training modules. Documentation of training will be maintained in the study coordinator's office. Agreeing to participate with the NCDR®, an institution also agrees to random site monitoring and/or audits.
2. Data Checks All patients who agree to participate in NEXUS outcomes registry and subsequent statistical analysis will experience a complete date audit for both outcomes assessments and NCDR® data elements. NCDR® has algorithm limits for both CathPCI® Registry and Afib Ablation ® Registry. All registry elements require abstraction form Meditech source documents. Reports are titled Cardiology Procedure Note and Electrophysiology Procedure Note for PCI and Afib ablation, respectively. Quality/outcome metrics will be sampled in paper form -the sources documents. Information will then be populated into excel for scoring. All paper forms will be maintained for the life of the study.
3. Data Dictionary Complete Data Dictionaries are provided by NCDR® with data element numbers and associated limits and acceptable values for both Cath PCI ® and Afib Ablation ® Registry.
4. Standard Operating Procedures A complete NEXUS Registry Protocol will be on site held in the Cardiovascular Innovation & Research Institute at Valley View Hospital along with all regulatory information, lab certifications, training documents, IRB documents, license agreements, analytic agreements and process maps for informed consent for outcomes research. Note NCDR® registries obtained a waiver for informed consent.
5. Sample Size Assessment The number of patients necessary to demonstrate an effect for outcomes after PCI with low-volume operators is 49.

   Presently, outcomes after surgical and/or endocardial ablation are being piloted to determine sample size for a study powered at 90%.
6. Missing Data Every attempt will be made to reach patients to ensure they are not lost to follow-up. Statistical consult recommends last observation carried forward for missing data.
7. Statistical Analysis Plan. For the primary analysis, the 6-month change in mean SAQ will be tested using a 1-sample upper 1-sided t-test. With 49 completers the t-test will have 90.4% power to detect an improvement in mean SAQ score of 10 points. A linear regression model will be used for the secondary analysis to investigate factors which are associated with the 6-month change (month 6 - baseline) in mean SAQ score. Factors which will be investigated for inclusion in the model include sex, age, physician American Society Anesthesiologists (ASA) class, physician volume, access site, and Charlson comorbidity index. An all-possible regressions approach will be used during the model building process in which all possible regression models are fit. The models will then be evaluated using Mallows' Cp statistic where models with values of Cp less than p (the number of parameters) will be considered as strong candidates for the final model. The final model will be selected after considering both results from the model selection process and subject matter knowledge. The regression analysis will have greater power than the t-test used in the sample size justification due to the reduction in variability of the outcome measure by including additional factors in a regression model. Additional analyses include [need to add specifics here]. All analyses will be conducted using SAS 9.4M4 or greater software (SAS Institute, Inc., Cary, NC, USA).

Morbidity / Complications will be reported included but not limited to bleeding at access site, hematoma, cardiac tamponade, vascular perforation, peripheral vascular injuries, post procedure hematoma, and mortality.

Statistical Analysis Plan with Respect to Surgical and/ or Endocardial Ablation for Afib

This outcomes registry is in its early pilot analysis for Afib and hypothesis generating. For the primary analysis, the six-month change in mean AFEQT scores will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Candidates will be included in the study only if all the following conditions are met:

1. Age >18 years
2. The subject has been informed of the nature of the study, agrees to its provisions, is able to comprehend, and has provided informed consent.
3. The subject is available for follow-up.
4. The subject has a diagnosis of coronary artery disease or Afib.

Exclusion Criteria:

Candidates will be excluded from the study if any of the following conditions are present:

1. Failure and / or inability and / or unwillingness to provide informed consent.
2. Likely problems, in the judgement of the investigators, with maintaining follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All comers outcomes registry
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Atrial Fibrillation Effect on Quality -of-Life (AFEQT) questionnaire at designated follow-up intervals | Initial Analysis at baseline (administered pre-AF intervention) to follow-up intervals at 6 months and then annually thereafter up to 10 years
  The AFEQT is a validated disease specific questionnaire used for assessing clinical disease impact on ADLs, emotional status, satisfaction with treatment and quality of life.
Change from baseline in Veterans Rand (VR) 12 | Initial analysis at baseline (administered pre-AF intervention) to follow-up intervals at 6 months and annually thereafter up to 10 years
  The VR 12 is a 12-item health survey, validated quality of life questionnaire- open source
Number of patients that experience a re-admit status post intervention | Within 90 days post intervention
  The number of patients that are re-admitted with a Serious Adverse Event (SAE) or Adverse Event (AE) as a result of their index procedure

SECONDARY OUTCOMES:
Number of patients that are in sinus rhythm post AF intervention | Assessed 6 months post procedure and annually thereafter
  Number of patients that are in sinus rhythm as evidenced by by a Holter monitor 6 month and one year after index procedure
number of patients on anti-arrhythmic agents post intervention | After 3 months post intervention /ablation known as blanking period and measured annually thereafter
  The number of patients after an ablative strategy that require anti-arrhythmic medicines to maintain sinus rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Laws, MD, Principal Investigator — Valley View Hospital
Locations (1):
- Valley View Hospital, Glenwood Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No